CLINICAL TRIAL: NCT02239770
Title: Pharmacokinetics of Nicotine Film in Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Patricia Sue Grigson, Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 00000873
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Results first posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Smoking Cessation
Keywords: Nicotine; Random Delivery; Smoking Cessation; Plasma Nicotine; Oral Film
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 0 mg Nicotine Film (Placebo Comparator): In Part 1, 4 participants will be allocated to this arm and receive one placebo nicotine film.
  Interventions: Drug: Placebo Nicotine Film
- 2 mg Nicotine Film (Experimental): In Part 1, 4 participants will be allocated to this arm and receive one 2 mg nicotine film.
  Interventions: Drug: Nicotine Film
- 4 mg Nicotine Film (Experimental): In Part 1, 4 participants will be allocated to this arm and receive one 4 mg nicotine film.
  Interventions: Drug: Nicotine Film
- 0, 0, 0, 0mg Nicotine Film Regimen (Placebo Comparator): In Part 2, 4 participants will be allocated to this arm and receive one nicotine film every 3 hours (for a total of 4 films over 12 hours) in the following order: 0, 0, 0, 0 mg.
  Interventions: Drug: Placebo Nicotine Film
- 2, 2, 2, 2mg Nicotine Film Regimen (Experimental): In Part 2, 4 participants will be allocated to this arm and receive one nicotine film every 3 hours (for a total of 4 films over 12 hours) in the following order: 2, 2, 2, 2 mg.
  Interventions: Drug: Nicotine Film
- 4, 4, 0, 4mg Nicotine Film Regimen (Experimental): In Part 2, 4 participants will be allocated to this arm and receive one nicotine film every 3 hours (for a total of 4 films over 12 hours) in the following order: 4, 4, 0, 4 mg.
  Interventions: Drug: Nicotine Film

INTERVENTIONS:
Drug: Nicotine Film — Nicotine orally dissolving films (ODF) are films containing nicotine (0, 2, or 4 mg). The active pharmaceutical ingredient in Nicotine ODF is nicotine polacrilex (20%, USP). The film used in Nicotine ODF has a muco-adhesive property, i.e. it can adhere to the oral mucosa and allow the drug to be absorbed through oral mucosa. After placement in the oral cavity, nicotine ODF dissolves over a 5-10 minute period.The unit-dose dosage is in the form of 1 in x 1 in square and weighs about 100 mg. Nicotine films are not available in the United States in a non-investigational setting.
  Arms: 2 mg Nicotine Film; 2, 2, 2, 2mg Nicotine Film Regimen; 4 mg Nicotine Film; 4, 4, 0, 4mg Nicotine Film Regimen
Drug: Placebo Nicotine Film — Nicotine orally dissolving films (ODF) are films containing nicotine (0, 2, or 4 mg). The active pharmaceutical ingredient in Nicotine ODF is nicotine polacrilex (20%, USP). The film used in Nicotine ODF has a muco-adhesive property, i.e. it can adhere to the oral mucosa and allow the drug to be absorbed through oral mucosa. After placement in the oral cavity, nicotine ODF dissolves over a 5-10 minute period.The unit-dose dosage is in the form of 1 in x 1 in square and weighs about 100 mg. Nicotine films are not available in the United States in a non-investigational setting.
  Arms: 0 mg Nicotine Film; 0, 0, 0, 0mg Nicotine Film Regimen

SUMMARY:
The objective of this study is to test the effect of a range of doses of a novel nicotine film on plasma nicotine levels, expired carbon monoxide and, via a questionnaire, subjective ratings of the film and side effects. The nicotine film is not part of standard of care and is not available in a non-investigational setting. The investigators hypothesize that plasma nicotine levels will be in keeping with those induced by other oral nicotine replacement therapies (NRTs) and by the smoking of a cigarette. Thus, the investigators predict that random delivery of nicotine via the oral film will be safe and well-tolerated by the human subjects.

DETAILED DESCRIPTION:
Briefly, this will be a two-part pharmacokinetic study, each part involving 12 participants.

In Part 1, 4 volunteer smokers (both male, and female) each will each abstain from all tobacco/nicotine products for 16 hours before attending the Penn State Clinical Research Center for the measurement of the blood nicotine pharmacokinetic response to a randomly allocated dose of either (a) 0mg, (b) 2mg or (c) 4mg oral nicotine film. A trained nurse will implant an intravenous indwelling catheter in each participant, through which they will provide a baseline blood sample after 16 hours of abstinence, confirmed by an exhaled carbon-monoxide < 6 ppm, and then will place a nicotine film in their mouth and have blood drawn every 10 minutes for the next 60 minutes, and then every 30 minutes for the next 2 hours plus one blood draw one minute after the film dissolves (11 blood draws in all over 3 hours after using the nicotine film). Subjective measures of (a) nicotine withdrawal and craving and (b) potential nicotine effects, including symptoms of nicotine intoxication, will be recorded at scheduled intervals through the study visit, and blood pressure and heart rate will be measured every 30 minutes. The investigators expect to find peak blood nicotine concentrations of around 3-4 ng/ml and 5-6 ng/ml from each of the two active doses of nicotine film, with the peak occurring approximately 30 minutes after film administration, and the level having dropped by at least half by 2 hours later. These peak blood nicotine levels are all within the range that a smoker might obtain after smoking a single cigarette. Upon completion of all blood draws, a trained nurse will remove the catheter and treat the puncture wound. The participant will receive $120 for this visit.

In Part 2, 12 participants will again attend the Penn State Clinical Research Center after 16 hours of abstinence, confirmed by an exhaled carbon monoxide < 12 ppm. On this visit participants will consume repeated doses of nicotine films intended to mimic the patterns of delivery that will be used in smoking cessation study 2 and fMRI study 3. The primary issue here is to determine peak blood nicotine concentrations and safety resulting from (a) the highest dose schedule that could be used in study 2 and 3, (b) the steady state levels produced by repeated administration of the 2mg nicotine film, and (c) to compare the subjective effects to placebo. In order to mimic the most aggressive dosing schedule possible in the "random nicotine" arm of study 2 and 3, the investigators will assess blood nicotine, subjective and basic cardiovascular responses to consuming nicotine film every 3 hours beginning at 8:00 a.m. on the following schedule: 4mg, 4mg, 0mg, 4mg.

All 12 participants will attend after 16 hours nicotine abstinence. 4 subjects each will be randomly allocated to consume 4 films over 12 hours in each of the following orders (a) 0,0,0,0 mg (b) 2,2,2,2 or (c) 4,4,0,4. A blood sample will be drawn at baseline prior to each film administration, and then at 30, 60 and 120 minutes after each film administration as well as one minute after film dissolution (20 blood draws in total), with heart rate and BP being assessed every 30 minutes. Nicotine has a half-life of approximately 2 hours, so the investigators expect that with 3-hourly administration there will not be much build-up of nicotine levels and these levels will be on the low end of the typical levels experienced by smokers every day. The participants will each receive $240 for this visit.

At clinic visits, in addition to providing blood samples for measurement of plasma nicotine concentration, participants will be asked to complete a battery of survey instruments assessing subjective effects (e.g. withdrawal and craving) and physical symptoms (e.g. dizziness and nausea) that could be caused by either nicotine withdrawal or nicotine exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 - 55
2. Smoke >9 cigarettes/day for at least the past 12 months
3. Able to understand and consent to study procedures
4. Able to read and write in English
5. Exhaled Carbon Monoxide <12 ppm at in-person screening

Exclusion Criteria:

1. Unstable or significant medical conditions and conditions such as elevated blood pressure (Systolic >140 mm Hg or diastolic >90mm Hg at baseline), COPD and those that are likely to affect biomarker data such as kidney or liver disease.
2. Individuals with sodium-restricted diet, heart disease, recent heart attack, irregular heartbeat, stomach ulcers, or diabetes as well as those taking prescription medications for depression or asthma as indicated under "Warnings" section on FDA approved NRT Drug Facts Label.
3. More than weekly use in the past 3 months of illegal drugs or prescription drugs that are not being used for medically prescribed purposes or inpatient treatment for these in the past 6 months.
4. Use of non-cigarette nicotine delivery product in the prior week (including cigars, pipes, chew, snus, hookah, electronic cigarette and marijuana mixed with tobacco).
5. Use of an FDA approved cessation medication in past week (any NRT, Chantix, Wellbutrin)
6. Women who are pregnant (verified by urine pregnancy test at visit), trying to become pregnant (not using a medically acceptable form of birth control for at least one month prior to visit i.e., oral contraceptives, intrauterine device, double barrier), or nursing.
7. Uncontrolled serious psychiatric illness or inpatient treatment in the past 6 months.
8. Unwillingness to provide blood samples or history of repeatedly fainting during blood draws
9. Any previous adverse reaction to NRT.
10. Any other condition, serious illness, or situation that would, in the investigator's opinion, make it unlikely that the participant could comply with the study protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia S. Grigson, Ph.D., Principal Investigator — Penn State College of Medicine; Jonathan A Foulds, Ph.D., Principal Investigator — Penn State College of Medicine; Christopher N Sciamanna, MD, MPH, Study Director — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine/Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In-person screening procedures included a review of medications and medical history, an assessment of drug use, a blood pressure measurement, a urine pregnancy test (if applicable), and an exhaled CO measurement to confirm prior 16 hour smoking abstinence. Those who did not satisfy inclusion criteria were excluded prior to randomization.
Groups:
- 0 mg Nicotine Film: In Part 1, 4 participants were allocated to this arm and received one placebo nicotine film.
  Placebo Nicotine Film: Nicotine orally dissolving films (ODF) are films containing nicotine (0, 2, or 4 mg). The active pharmaceutical ingredient in Nicotine ODF is nicotine polacrilex (20%, USP). The film used in Nicotine ODF has a muco-adhesive property, i.e. it can adhere to the oral mucosa and allow the drug to be absorbed through oral mucosa. After placement in the oral cavity, nicotine ODF dissolves over a 5-10 minute period.The unit-dose dosage is in the form of 1 in x 1 in square and weighs about 100 mg. Nicotine films are not available in the United States in a non-investigational setting.
- 2 mg Nicotine Film: In Part 1, 4 participants were allocated to this arm and received one 2mg nicotine film.
  Nicotine Film: Nicotine orally dissolving films (ODF) are films containing nicotine (0, 2, or 4 mg). The active pharmaceutical ingredient in Nicotine ODF is nicotine polacrilex (20%, USP). The film used in Nicotine ODF has a muco-adhesive property, i.e. it can adhere to the oral mucosa and allow the drug to be absorbed through oral mucosa. After placement in the oral cavity, nicotine ODF dissolves over a 5-10 minute period.The unit-dose dosage is in the form of 1 in x 1 in square and weighs about 100 mg. Nicotine films are not available in the United States in a non-investigational setting.
- 4 mg Nicotine Film: In Part 1, 4 participants were allocated to this arm and received one 4mg nicotine film.
  Nicotine Film: Nicotine orally dissolving films (ODF) are films containing nicotine (0, 2, or 4 mg). The active pharmaceutical ingredient in Nicotine ODF is nicotine polacrilex (20%, USP). The film used in Nicotine ODF has a muco-adhesive property, i.e. it can adhere to the oral mucosa and allow the drug to be absorbed through oral mucosa. After placement in the oral cavity, nicotine ODF dissolves over a 5-10 minute period.The unit-dose dosage is in the form of 1 in x 1 in square and weighs about 100 mg. Nicotine films are not available in the United States in a non-investigational setting.
- 0, 0, 0, 0mg Nicotine Film Regimen: In Part 2, 4 participants were allocated to this arm and received one nicotine film every 3 hours (for a total of 4 films over 12 hours) in the following order: 0, 0, 0, 0 mg.
  Placebo Nicotine Film: Nicotine orally dissolving films (ODF) are films containing nicotine (0, 2, or 4 mg). The active pharmaceutical ingredient in Nicotine ODF is nicotine polacrilex (20%, USP). The film used in Nicotine ODF has a muco-adhesive property, i.e. it can adhere to the oral mucosa and allow the drug to be absorbed through oral mucosa. After placement in the oral cavity, nicotine ODF dissolves over a 5-10 minute period.The unit-dose dosage is in the form of 1 in x 1 in square and weighs about 100 mg. Nicotine films are not available in the United States in a non-investigational setting.
- 2, 2, 2, 2mg Nicotine Film Regimen: In Part 2, 4 participants were allocated to this arm and received one nicotine film every 3 hours (for a total of 4 films over 12 hours) in the following order: 2, 2, 2, 2 mg.
  Nicotine Film: Nicotine orally dissolving films (ODF) are films containing nicotine (0, 2, or 4 mg). The active pharmaceutical ingredient in Nicotine ODF is nicotine polacrilex (20%, USP). The film used in Nicotine ODF has a muco-adhesive property, i.e. it can adhere to the oral mucosa and allow the drug to be absorbed through oral mucosa. After placement in the oral cavity, nicotine ODF dissolves over a 5-10 minute period.The unit-dose dosage is in the form of 1 in x 1 in square and weighs about 100 mg. Nicotine films are not available in the United States in a non-investigational setting.
- 4, 4, 0, 4mg Nicotine Film Regimen: In Part 2, 4 participants were allocated to this arm and received one nicotine film every 3 hours (for a total of 4 films over 12 hours) in the following order: 4, 4, 0, 4 mg.
  Nicotine Film: Nicotine orally dissolving films (ODF) are films containing nicotine (0, 2, or 4 mg). The active pharmaceutical ingredient in Nicotine ODF is nicotine polacrilex (20%, USP). The film used in Nicotine ODF has a muco-adhesive property, i.e. it can adhere to the oral mucosa and allow the drug to be absorbed through oral mucosa. After placement in the oral cavity, nicotine ODF dissolves over a 5-10 minute period.The unit-dose dosage is in the form of 1 in x 1 in square and weighs about 100 mg. Nicotine films are not available in the United States in a non-investigational setting.
Period: Part 1
Arm/Group | 0 mg Nicotine Film | 2 mg Nicotine Film | 4 mg Nicotine Film | 0, 0, 0, 0mg Nicotine Film Regimen | 2, 2, 2, 2mg Nicotine Film Regimen | 4, 4, 0, 4mg Nicotine Film Regimen
Started | 4 | 4 | 4 | 0 | 0 | 0
Completed | 4 | 4 | 4 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | 0 mg Nicotine Film | 2 mg Nicotine Film | 4 mg Nicotine Film | 0, 0, 0, 0mg Nicotine Film Regimen | 2, 2, 2, 2mg Nicotine Film Regimen | 4, 4, 0, 4mg Nicotine Film Regimen
Started | 0 | 0 | 0 | 4 | 4 | 4
Completed | 0 | 0 | 0 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 2 mg Nicotine Film: In Part 1, 4 participants were allocated to this arm and received one 2 mg nicotine film.
  Nicotine Film: Nicotine orally dissolving films (ODF) are films containing nicotine (0, 2, or 4 mg). The active pharmaceutical ingredient in Nicotine ODF is nicotine polacrilex (20%, USP). The film used in Nicotine ODF has a muco-adhesive property, i.e. it can adhere to the oral mucosa and allow the drug to be absorbed through oral mucosa. After placement in the oral cavity, nicotine ODF dissolves over a 5-10 minute period.The unit-dose dosage is in the form of 1 in x 1 in square and weighs about 100 mg. Nicotine films are not available in the United States in a non-investigational setting.
- 4 mg Nicotine Film: In Part 1, 4 participants were allocated to this arm and received one 4 mg nicotine film.
  Nicotine Film: Nicotine orally dissolving films (ODF) are films containing nicotine (0, 2, or 4 mg). The active pharmaceutical ingredient in Nicotine ODF is nicotine polacrilex (20%, USP). The film used in Nicotine ODF has a muco-adhesive property, i.e. it can adhere to the oral mucosa and allow the drug to be absorbed through oral mucosa. After placement in the oral cavity, nicotine ODF dissolves over a 5-10 minute period.The unit-dose dosage is in the form of 1 in x 1 in square and weighs about 100 mg. Nicotine films are not available in the United States in a non-investigational setting.
- Total: Total of all reporting groups
Arm/Group | 0 mg Nicotine Film | 2 mg Nicotine Film | 4 mg Nicotine Film | 0, 0, 0, 0mg Nicotine Film Regimen | 2, 2, 2, 2mg Nicotine Film Regimen | 4, 4, 0, 4mg Nicotine Film Regimen | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (11.8) | 40.8 (13.6) | 31.8 (11.0) | 44.8 (6.5) | 36.0 (12.3) | 37.5 (14.7) | 38.0 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 3 | 1 | 1 | 10
  Male | 2 | 2 | 3 | 1 | 3 | 3 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian/white | 4 | 3 | 4 | 2 | 2 | 2 | 17
  Race: African American/black | 0 | 1 | 0 | 1 | 1 | 2 | 5
  Race: Other | 0 | 0 | 0 | 1 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 4 | 4 | 4 | 4 | 4 | 24
Less than a college degree [Count of Participants; unit: Participants] | 3 | 3 | 2 | 2 | 2 | 3 | 15
Cigarettes smoked per day [Mean (Standard Deviation); unit: cigarettes per day] | 20 (8.0) | 20 (0.0) | 14 (3.0) | 18.8 (5.1) | 18.5 (8.6) | 14.8 (6.3) | 17.7 (5.8)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.7 (6.4) | 30.1 (10.0) | 27.2 (2.1) | 28.7 (3.5) | 26.9 (4.2) | 27.4 (5.3) | 28.2 (5.3)
Exhaled carbon monoxide [Mean (Standard Deviation); unit: parts per million] | 5.0 (3.0) | 6.0 (2.0) | 4.0 (3.0) | 7.0 (2.2) | 6.3 (3.3) | 5.8 (3.2) | 5.6 (2.8)
Penn State Cigarette Dependence Index Total Score [Mean (Standard Deviation); unit: units on a scale] — The total score of the Penn State Cigarette Dependence Index can range from 0 (no dependence/better outcome) to 20 (high dependence/worse outcome).
  A score of 0 to 3 indicates no dependence on cigarettes. A score of 4 to 8 indicates low dependence on cigarettes. A score of 9 to 12 indicates medium dependence on cigarettes. A score of 13 or higher indicates a high dependence on cigarettes.
  units on a scale | 14 (3.0) | 12 (1.0) | 11 (2.0) | 11.8 (2.9) | 10.8 (3.8) | 11.0 (2.2) | 11.6 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Nicotine Concentrations Following Ingestion of a Single (Phase 1) or Repeated (Phase 2) Doses of Nicotine Film
Description: In Phase 1, a trained nurse will implant an intravenous (IV) indwelling catheter in each participant. Participants will place a film containing zero, 2, or 4 mg of nicotine in their mouths and blood will be drawn every 10 minutes thereafter for the next 60 minutes, and then every 30 minutes for the next 2 hours (11 blood draws in all over 3 hours after using the nicotine film).
  In Phase 2, all 12 participants will receive an IV catheter and randomly allocated to consume 4 films over 12 hours in each of the following orders (a) 0,0,0,0 mg (b) 2,2,2,2 or (c) 4,4,0,4. A blood sample will be drawn at baseline prior to each film administration, and then at 30, 45, 60 and 120 minutes after each film administration and when the film is reported dissolved (20 blood draws in total).
Time Frame: 10 min - 12 hours
Population: Because the placebo nicotine film does not deliver any nicotine to the blood, peak plasma nicotine levels cannot be observed in the 0 mg Nicotine Film arm (Part 1) and 0, 0, 0, 0 mg Nicotine Film Regimen (Part 2).
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | 0 mg Nicotine Film | 2 mg Nicotine Film | 4 mg Nicotine Film | 0, 0, 0, 0mg Nicotine Film Regimen | 2, 2, 2, 2mg Nicotine Film Regimen | 4, 4, 0, 4mg Nicotine Film Regimen
Number analyzed (Participants) | 0 | 4 | 4 | 0 | 4 | 4
ng/mL |  | 5.78 [3.7 to 8.2] | 20.5 [15.9 to 31.0] |  | 8.71 [5.25 to 15.5] | 8.80 [3.96 to 14.86]

2. Secondary Outcome: Questionnaire of Smoking Urges-Brief Mean Total Score by Dose Group
Description: The Questionnaire of Smoking Urges-Brief (QSU-Brief) with a possible total score range of 10 to 70 was used to measure cigarette craving at baseline and at several points throughout the study visit for each participant. A score of 10 on this scale indicates very low cigarette craving, while a score of 70 indicates very high cigarette craving.
  Part 1: The QSU-Brief was measured at baseline and at 15, 35, 55, 80, 140, and 200 minutes post film administration.
  Part 2: The QSU-Brief was measured at baseline and at 50, 110, 230, 290, 410, 470, 590, and 690 minutes post FIRST film administration.
Time Frame: Part 1: The QSU-Brief was measured at baseline and at 15, 35, 55, 80, 140, and 200 minutes post film administration. Part 2: The QSU-Brief was measured at baseline and at 50, 110, 230, 290, 410, 470, 590, and 690 minutes post FIRST film administration.
Population: This was a two part study. Participants in Part 1 and Part 2 were not assessed on the QSU-Brief measure at the same time intervals due to the differing study visit structures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0 mg Nicotine Film | 2 mg Nicotine Film | 4 mg Nicotine Film | 0, 0, 0, 0mg Nicotine Film Regimen | 2, 2, 2, 2mg Nicotine Film Regimen | 4, 4, 0, 4mg Nicotine Film Regimen
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
score on a scale
  0 minute | 56.3 (8.4) | 35.0 (16.4) | 46.0 (8.3) | 51.8 (19.3) | 46.3 (23.0) | 39.3 (15.6)
  15 minutes: number analyzed (Participants) | 4 | 4 | 4 | 0 | 0 | 0
  15 minutes | 43.3 (14.2) | 22.8 (8.5) | 26.5 (7.1) |  |  |
  35 minutes: number analyzed (Participants) | 4 | 4 | 4 | 0 | 0 | 0
  35 minutes | 35.0 (10.8) | 23.8 (12) | 22.5 (9.9) |  |  |
  50 minutes: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 4
  50 minutes |  |  |  | 40.5 (15.9) | 30.8 (15.4) | 25.5 (15.6)
  55 minutes: number analyzed (Participants) | 4 | 4 | 4 | 0 | 0 | 0
  55 minutes | 29.8 (14.7) | 18.0 (5.7) | 19.0 (9.2) |  |  |
  80 minutes: number analyzed (Participants) | 4 | 4 | 4 | 0 | 0 | 0
  80 minutes | 31.5 (16.8) | 16.8 (4.8) | 24.3 (9.7) |  |  |
  110 minutes: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 4
  110 minutes |  |  |  | 39.5 (3.8) | 31.5 (16.0) | 27.0 (15.6)
  140 minutes: number analyzed (Participants) | 4 | 4 | 4 | 0 | 0 | 0
  140 minutes | 36.0 (19.4) | 16.5 (3.9) | 22.0 (10.4) |  |  |
  200 minutes: number analyzed (Participants) | 4 | 4 | 4 | 0 | 0 | 0
  200 minutes | 37.3 (25.4) | 18.3 (6.4) | 26.0 (13.3) |  |  |
  230 minutes: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 4
  230 minutes |  |  |  | 35.5 (11.4) | 32.0 (21.4) | 24.0 (13.0)
  290 minutes: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 4
  290 minutes |  |  |  | 42.3 (11.3) | 34.5 (23.9) | 28.0 (20.6)
  410 minutes: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 4
  410 minutes |  |  |  | 36.0 (18.0) | 29.0 (19.7) | 28.5 (14.1)
  470 minutes: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 4
  470 minutes |  |  |  | 32.8 (17.2) | 29.3 (18.9) | 31.3 (18.2)
  590 minutes: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 4
  590 minutes |  |  |  | 29.8 (14.4) | 36.0 (27.1) | 23.5 (18.4)
  690 minutes: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 4
  690 minutes |  |  |  | 30.3 (16.6) | 31.5 (20.9) | 26.8 (18.8)

3. Secondary Outcome: Mean Systolic Blood Pressure
Description: Systolic blood pressure was measured using an electronic sphygmomanometer just prior to film administration and at every 30 minutes after film administration for the duration of each study visit.
Time Frame: Part 1: Systolic blood pressure was measured at baseline and at every 30 minutes, up to 180 minutes post film administration. Part 2: Systolic blood pressure was measured at baseline and at every 30 minutes, up to 660 minutes post film administration.
Population: Participants in Part 1 of the study were not assessed past 180 minutes post film administration, as this was the extent of the study visit.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 0 mg Nicotine Film | 2 mg Nicotine Film | 4 mg Nicotine Film | 0, 0, 0, 0mg Nicotine Film Regimen | 2, 2, 2, 2mg Nicotine Film Regimen | 4, 4, 0, 4mg Nicotine Film Regimen
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
mmHg
  Baseline | 118.0 (12.8) | 115.8 (17.3) | 118.0 (17.1) | 114.8 (12.2) | 123.0 (8.8) | 125.5 (5.8)
  30 minutes | 120.5 (15.8) | 110.8 (13.6) | 125.8 (11.4) | 110.3 (10.8) | 128.8 (6.8) | 129.5 (9.9)
  60 minutes | 121.8 (17.0) | 117.8 (14.5) | 118.5 (20.0) | 108.3 (12.8) | 129.5 (5.5) | 131.3 (8.3)
  90 minutes | 120.8 (16.1) | 116.0 (14.1) | 120.3 (11.8) | 108.8 (9.2) | 121.0 (11.5) | 128.3 (17.9)
  120 minutes | 118.5 (10.5) | 114.5 (15.9) | 115.3 (12.5) | 110.3 (2.5) | 125.8 (8.7) | 127.5 (3.1)
  150 minutes | 116.3 (10.6) | 110.5 (14.5) | 113.3 (16.1) | 99.0 (8.0) | 126.5 (12.2) | 123.0 (10.9)
  180 minutes | 114.3 (4.1) | 118.8 (14.8) | 115.5 (13.8) | 104.5 (3.1) | 127.0 (7.3) | 122.8 (10.4)
  210 minutes: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 4
  210 minutes |  |  |  | 104.8 (7.2) | 124.0 (11.3) | 125.5 (9.4)
  240 minutes: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 4
  240 minutes |  |  |  | 116.0 (8.9) | 127.8 (13.7) | 122.8 (4.5)
  270 minutes: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 4
  270 minutes |  |  |  | 115.0 (8.9) | 129.8 (11.0) | 122.5 (6.5)
  300 minutes: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 4
  300 minutes |  |  |  | 109.3 (8.0) | 122.0 (14.3) | 124.8 (3.3)
  330 minutes: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 4
  330 minutes |  |  |  | 109.0 (5.9) | 124.3 (6.7) | 120.0 (3.6)
  360 minutes: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 4
  360 minutes |  |  |  | 109.0 (8.8) | 120.5 (15.6) | 125.8 (4.1)
  390 minutes: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 4
  390 minutes |  |  |  | 106.8 (11.0) | 124.0 (5.4) | 123.3 (3.5)
  420 minutes: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 4
  420 minutes |  |  |  | 115.5 (6.9) | 126.5 (11.4) | 124.8 (14.3)
  450 minutes: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 4
  450 minutes |  |  |  | 112.8 (9.7) | 131.3 (3.3) | 123.8 (13.8)
  480 minutes: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 4
  480 minutes |  |  |  | 107.5 (5.2) | 127.8 (11.4) | 121.3 (6.3)
  510 minutes: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 4
  510 minutes |  |  |  | 111.3 (5.6) | 124.5 (7.0) | 122.8 (7.6)
  540 minutes: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 4
  540 minutes |  |  |  | 113.8 (11.8) | 129.0 (8.0) | 115.5 (5.0)
  570 minutes: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 4
  570 minutes |  |  |  | 151.0 (11.3) | 129.3 (10.2) | 115.5 (3.8)
  600 minutes: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 4
  600 minutes |  |  |  | 111.3 (9.1) | 125.0 (12.9) | 123.0 (8.3)
  630 minutes: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 4
  630 minutes |  |  |  | 108.3 (14.5) | 134.8 (7.0) | 121.5 (1.7)
  660 minutes: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 4
  660 minutes |  |  |  | 109.5 (15.9) | 134.5 (7.8) | 121.3 (3.9)

ADVERSE EVENTS:
Time Frame: In Part 1, adverse event data were collected throughout the entirety of the study visit lasting approximately 4 hours in length. In Part 2, adverse event data were collected throughout the entirety of the study visit lasting approximately 12 hours in length.
Arm/Group | 0 mg Nicotine Film | 2 mg Nicotine Film | 4 mg Nicotine Film | 0, 0, 0, 0mg Nicotine Film Regimen | 2, 2, 2, 2mg Nicotine Film Regimen | 4, 4, 0, 4mg Nicotine Film Regimen
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/4 | 1/4 | 2/4 | 0/4 | 3/4 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0 mg Nicotine Film (N=4) | 2 mg Nicotine Film (N=4) | 4 mg Nicotine Film (N=4) | 0, 0, 0, 0mg Nicotine Film Regimen (N=4) | 2, 2, 2, 2mg Nicotine Film Regimen (N=4) | 4, 4, 0, 4mg Nicotine Film Regimen (N=4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT02239770/Prot_SAP_000.pdf